CLINICAL TRIAL: NCT00000321
Title: Methamphetamine Abuse Pharmacology in Patients With AIDS
Brief Title: Methamphetamine Abuse Treatment in Patients With AIDS - 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Friends Research Institute, Inc. (Other)
Purpose: Treatment
Other Study IDs: NIDA-10643-1; R01-10643-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1996-10

CONDITIONS: Substance-Related Disorders
Keywords: methamphetamine dependence
MeSH Terms: conditions — Substance-Related Disorders | interventions — Desipramine

INTERVENTIONS:
Drug: Desipramine

SUMMARY:
The purpose of this study is to evaluate the efficacy of desipramine, sertraline, and placebo on methamphetamine dependent gay men with AIDS.

ELIGIBILITY:
Please contact site for information.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 1996-10; Study Completion 2001-12

PRIMARY OUTCOMES:
Craving
Retention
Depression
Methamphetamine use
Anxiety and Depression
ASI Scales (7)
AIDS medical care engagement
High risk sexual behaviors
Mood indicators

CONTACTS AND LOCATIONS:
Overall Officials: Frank Gawin, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States